CLINICAL TRIAL: NCT03562702
Title: Comparative Study Between the Oral Rehydration Product, Speedlyte, With Lipophilic Absorption and IV Rehydration in Treatment of Children With Gastroenteritis in a Pediatric Emergency Department
Brief Title: Comparing Speedlyte and IV Rehydration Treating Children With Gastroenteritis in a Pediatric Emergency Department (ED)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Access to Speedlyte Product no longer available.
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Collaborators: Einsoff Biohealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCH09017
Record Dates: First submitted 2018-04-19; First posted 2018-06-19 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Dehydration; Acute Gastroenteritis
Keywords: vomiting; diarrhea
MeSH Terms: conditions — Dehydration; Vomiting; Diarrhea | interventions — Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The assignment of treatment will be concealed from research team members involved in recruiting patients by using sealed, sequentially numbered, opaque envelopes containing the type of rehydration treatment to be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard IV Rehydration Therapy (Active Comparator): Patients randomized into the IV rehydration group will receive a Normal Saline bolus of IVF (usually 20 mL/kg) which is the standard therapy up to 24 hrs or as needed depending on patient's weight
  Interventions: Other: Standard IV Rehydration Therapy; Other: Oral Rehydration Therapy (ORT)
- Oral Rehydration Therapy (ORT) (Experimental): Patients randomized into the oral rehydration group will receive the oral Speedlyte product instead of the IV rehydration therapy.
  Interventions: Other: Standard IV Rehydration Therapy; Other: Oral Rehydration Therapy (ORT)

INTERVENTIONS:
Other: Standard IV Rehydration Therapy — IV rehydration group receiving a Normal Saline bolus of IVF (usually 20 ml/kg)
Other: Oral Rehydration Therapy (ORT) — Speedlyte oral solution as rehydration therapy based on participant's weight (10 m/l kg over one hour). Total of 150 ml/kg over 24 hours prior to discharge

SUMMARY:
To compare length of stay (LOS) of pediatric patients in a pediatric emergency room presenting with Gastroenteritis treated with IV rehydration versus oral Speedlyte rehydration.

DETAILED DESCRIPTION:
Gastroenteritis leading to dehydration is very commonly encountered in the pediatric emergency room setting. Oral rehydration therapy (ORT) is the first line therapy recommended by the American Academy of Pediatrics but is seldom used compared to intravenous therapy (IVT). ORT has many advantages including less traumatic to the patient, can be administered by mouth, can be administered at home and less costly compared to IVT. Furthermore, intravenous fluids may present several complications with IV placement such as infiltration, hematoma, air embolism, phlebitis, extravascular injection, intraarterial injection, etc. Speedlyte is a new oral rehydration product with lipophilic absorption which allows for electrolytes to be more readily absorbed compared to other oral rehydration solutions. The liposome encapsulates the salty molecules which is thought to decrease the negative salty taste associated with oral rehydration solutions. In addition, the encapsulation of electrolytes allows for more molecules to be delivered past the stomach acids and absorbed into the body under higher bioavailability due to the lipid shell.

Participants will be randomized into two rehydration groups. One group will receive oral rehydration with the Speedlyte product, the amount will be based on the participant's weight. The other group will receive intravenous rehydration with a normal saline bolus per physician practice, usually in the amount of 20 mL/kg. These interventions can be incorporated into the emergency room practice without undue expense to the setting or placing excessive demands on nursing time as these practices are standard of care in many rehydration cases.

ELIGIBILITY:
Inclusion Criteria:

* 6 mths to 18 years;
* Signs and symptoms of dehydration for less than a week
* Diagnosis of acute gastroenteritis, dehydration, vomiting, and/or diarrhea;
* Patient able to drink from bottle and/or cup;
* Per clinician's judgment, patient needs rehydration with IV solution.

Exclusion Criteria:

* Chronic disease that includes but not limited to TB, HIV, congenital heart disease with hemodynamic consequences, metabolic disease, cerebral palsy, adrenal hyperplasia, renal tubular acidosis, and nephropathy;
* Vomiting due to head trauma;
* Severe hydration;
* Diabetic ketoacidosis;
* Bloody diarrhea;
* Diarrhea for more than a week;
* Malnutrition;
* Burns;
* Pneumonia;
* Meningitis;
* History of seizures;
* Absent bowel sounds;
* Not able to drink from bottle or cup;
* Previous allergic reaction to citrate or other food coloring particles/formulation;
* Parent/legal guardian refusing to participate.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Length of stay (LOS) | up to 24 hours
  Comparison of length of stay (LOS) in a pediatric emergency department in the treatment of acute gastroenteritis between the oral rehydration solution Speedlyte and intravenous rehydration.

SECONDARY OUTCOMES:
Adjunct Medication | up to 24 hours
  Number of adjunct medications given in the ED in both groups

OTHER OUTCOMES:
Time to initiation of therapy | up to 24 hours
  Time to initiation of therapy in each group
Number of patients that fail to rehydrate | up to 24 hours
  Obtain the number of patients that fail to rehydrate in each group. Oral requiring IV intervention, IV requiring further fluids and/or admission.
Hospitalization rate | up to 24 hours
  The rate of hospitalization for each group
Revisit rate in each group. | up to 24 hours
  The revisit rate for each group

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pena, MD, Principal Investigator — Nicklaus Children's Hospital
Locations (1):
- Nicklaus Children's Hospital f/k/a Miami Children's Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellemare S, Hartling L, Wiebe N, Russell K, Craig WR, McConnell D, Klassen TP. Oral rehydration versus intravenous therapy for treating dehydration due to gastroenteritis in children: a meta-analysis of randomised controlled trials. BMC Med. 2004 Apr 15;2:11. doi: 10.1186/1741-7015-2-11. PMID 15086953
- [Background] Spandorfer PR, Alessandrini EA, Joffe MD, Localio R, Shaw KN. Oral versus intravenous rehydration of moderately dehydrated children: a randomized, controlled trial. Pediatrics. 2005 Feb;115(2):295-301. doi: 10.1542/peds.2004-0245. PMID 15687435